CLINICAL TRIAL: NCT00352352
Title: Randomized Control Trial of Using Acupuncture In Children With Autistic Spectrum Disorder
Brief Title: Use of Acupuncture In Children With Autistic Spectrum Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3469296479554546
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2006-07-14 (Estimated); Status verified 1999-07

CONDITIONS: Autism; Autistic Disorder
Keywords: Traditional Chinese Medicine (TCM); Alternative Medicine (AM); Tongue Acupuncture (TAC); Autism Spectrum Disorder (ASD); Autism; Children
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

INTERVENTIONS:
Procedure: Tongue Acupuncture (Procedure)

SUMMARY:
This is a study of the efficacy of acupuncture in children with autism.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) or autism is a neurodevelopmental disorder with unknown etiology. ASD consisted of 3 core features: 1) disorder of language or communication; 2) disorder of social interaction; and 3) obsessive and stereotypic behavior.

Acupuncture had been practiced in China for over two millennia. In Traditional Chinese Acupuncture, nearly 400 acupoints on the body surface are interrelated to various functions. The approach in TCM, in sharp contrast to western medical concept, was a "holistic" approach with a philosophical background of balancing the "Yin-and-Yang". The main objective of TCM was to improve health of body and mind by deblocking the flow of "Qi" in the body. The pathophysiological basis of TCM aimed to improve "energy" or "body-flow" or "Qi" ["de-qui" in Chinese]. The effect of acupuncture was had been proven in animal and human studies to be due to direct neural stimulation, changes in neurotransmitters such as endorphin, immunological markers or endocrinological signals. Thus, acupuncture is especially effective in chronic disorders, especially neurological ones.

As there is no TCM concept of mental retardation or autism, we propose that ASD is part of the spectrum of the TCM concept of the "Four Delayed Syndrome" in children with "delay in motor skills, speech, hair and teeth eruption" according to TCM concept. Thus, we approach ASD according to TCM concept as part of the lower intelligence due to imbalance of "Heart meridian and Kidney meridian" (i.e. yin-yang imbalance) resulting in communication problem and "Liver meridian" (yin-yang imbalance) leading to behavioral problems.

Our objective is to use a different approach in looking at ASD and to assess the efficacy of TCM model in improving the functional status of these children. Specific acupoints corresponding to various organs and meridians were used for ASD. The organ and meridian concept in TCM model has been as a fundamental basis to improve the behavior, cognition and communicative ability in children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of ASD or autism was made according to the criteria of the 4th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and Autism Diagnostic Interview-Revised (ADI-R).
* The diagnosis of autism was made if it satisfied a score greater than 30 in the Childhood Autism Rating Scale (CARS).

Exclusion Criteria:

* Children with associated neurological disorders such as Tuberous Sclerosis, Fragile X Syndrome and epilepsy.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30

PRIMARY OUTCOMES:
Ritvo-Freeman Real Life Scale (RFRLS) was conducted on both groups before (Week 0) and after (Week 8) acupuncture.
Functional Independence Measure for children (WeeFIM) consists of 18 questions concerning on the Functional Independence Measure for children, which was conducted on both groups before (Week 0) and after (Week 8) acupuncture.
Parental Stress Index (PSI) consists of child domain, parent domain and a total domain, which was conducted on both groups before (Week 0) and after (Week 8) acupuncture.
Clinical Global Impression Scale (CGIS) is a measure in a Likert scale of 0 - 7, which was conducted on both groups before (Week 0) and after (Week 8) acupuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Wong Virginia, Principal Investigator — The University of Hong Kong
Locations (1):
- Duchess of Kent of Children Hospital, Hong Kong, Hong Kong